CLINICAL TRIAL: NCT01479894
Title: Genetic Analysis to Evaluate the Racial Difference in the Outcome of Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: Genomic Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: 133972
Record Dates: First submitted 2011-11-17; First posted 2011-11-28 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2015-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The Oncotype DX Colon Cancer Assay will be utilized to define the gene expression profile of the tumor tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sample Collection: This is an exploratory study utilizing archived tumor specimens and demographic and pathologic characteristics derived from the patient's medical charts. As such, all eligible patients must have a stored tumor specimen which can be accessed for analysis.

SUMMARY:
This is a retrospective genetic analysis of stored tumor tissue samples to evaluate the distribution of Recurrence Score® and gene groups of stage II colon cancer in African American (AA) and Caucasian individuals. Other covariant factors in the medical chart will be analyzed as well. Three institutions will contribute patients to this study with a total patient number goal of approximately 200 with approximately 100 being AA and approximately 100 being Caucasian. As enrollment in this study proceeds a Caucasian subject will be matched for every African American enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* Subjects must be AA or Caucasian.
* Subjects with pathologic stage II colon cancer; Irrespective of number of nodes examined.

Exclusion Criteria:

* Patients of races other than AA or Caucasian.
* No tumor block available from initial diagnosis.
* No tumor or very little tumor (<5% tumor present) in block as assessed by examination of the H&E slide by the Genomic Health, Inc (GHI) - designated pathologist.
* Tumor types other than adenocarcinoma NOS (not otherwise specified) and mucinous carcinoma as assessed by examination of the H&E slide by the GHI-designated pathologist.
* Insufficient RNA (<5 ng/μL or 300 ng) for RT-PCR (radiation therapy - pathologic complete response) analysis.
* Failure of assay to meet pre-specified quality control (QC) specifications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an exploratory study utilizing archived tumor specimens and demographic and pathologic characteristics derived from the patient's medical charts. As such, all eligible patients must have a stored tumor specimen which can be accessed for analysis.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Compare the prognosis of colon cancer patients compared to gene expression. | 1 year
  Compare the values of the Recurrence Score and expression levels of gene groups and individual genes between African Americans and Caucasians with Stage II colon cancer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States